CLINICAL TRIAL: NCT02157389
Title: Psychobiological Mechanisms of Placebo and Nocebo Effects in the Treatment of Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Prof Herta Flor, Prof. Dr. Herta Flor, Central Institute of Mental Health, Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Fl156/33-1_chrBP
Record Dates: First submitted 2014-06-03; First posted 2014-06-06 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Lower Back Pain; Healthy Control Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- placebo (Experimental): Administration of a pharmacological placebo (sodium chloride) via transdermal application to investigate the influence on pain perception in chronic back pain patients and to investigate the influence of attitude and experience with medication on the placebo effect
  Interventions: Other: Administration of a pharmacological placebo

INTERVENTIONS:
Other: Administration of a pharmacological placebo

SUMMARY:
Placebo and nocebo responses have mainly been studied in healthy humans for pharmacological rather than psychological interventions. Moreover, only few studies examined patients or tested how previous experience and attitudes affect placebo and nocebo responses. On the psychological level expectancy and classical conditioning have been identified as two primary mechanisms. Both seem to be important with classical conditioning potentially having more long-term effects and expectancy being more important in nocebo effects. There is some initial evidence from the investigators own research that patients may be more prone to these effects and the investigators have also shown that placebo effects may last up to several years after treatment. The investigators therefore examine previous attitudes to pharmacological interventions for chronic pain in patients with chronic back pain and subdivide them into groups with high of low belief in the respective treatment modality. The investigators then apply a pharmacological placebo and study the interaction between the prevailing attitude (implicit and explicit) and the placebo effect with respect to pain perception but also to neurobiological mechanisms using functional magnetic resonance imaging. In addition to expectancy, conditioning of placebo will be examined and the long-term effects of the intervention will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male and female human subjects with chronic back pain (chronic persistent and recurrent pain > 6 months)
* Age between 18 and 65
* Voluntary participation.

Exclusion Criteria:

* Acute or chronic somatic diseases and inflammatory, neuropathic or tumor-related pain
* Acute and chronic mental disorders according to DSM-IV (except for comorbid anxiety or depression, which are frequent in chronic pain)
* Insufficient German language skills
* Cognitive limitations
* Intake of opioid medication or tranquilizers
* Metal implants or electric implants that cannot be removed
* Pregnancy
* Claustrophobia
* History of epilepsy, brain trauma, or brain tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity and pain unpleasantness ratings after placebo intervention | immediatey to one week

SECONDARY OUTCOMES:
Changes in neuronal activity in response to painful stimulation after placebo administration | immediately
Changes in movement abilities after placebo administration | immediately to one week

CONTACTS AND LOCATIONS:
Overall Officials: Herta Flor, PhD, Principal Investigator — Medical Faculty Mannheim, Heidelberg University
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany